CLINICAL TRIAL: NCT03253861
Title: Risk Factors and Outcomes of Infected Pancreatic Necrosis: Retrospective Cohort of 148 Patients Admitted to the ICU for Acute Pancreatitis
Brief Title: PancRea: Risk Factors and Outcomes of Infected Pancreatic Necrosis
Acronym: PancRea
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC16_0126
Record Dates: First submitted 2017-08-16; First posted 2017-08-18 (Actual); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Acute Necrotizing Pancreatitis; Infection; Pancreatitis
Keywords: Acute necrotizing pancreatitis; Acute pancreatitis; Sepsis/complications; Infection; Organ Dysfunction Scores; Drainage; Catheters; Antibiotics; Multiresistant organism; Pancreatitis/complications; Pancreatitis/diagnosis; Pancreatitis/surgery; Pancreatitis/therapy; Pancreatitis, Acute Necrotizing/complications; Pancreatitis, Acute Necrotizing/surgery; Pancreatitis, Acute Necrotizing/therapy
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing; Infections; Pancreatitis; Sepsis; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control patients: patients without an infected pancreatic necrosis
  Interventions: Other: No intervention
- Case patients: patients with an infected pancreatic necrosis
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Severe acute pancreatitis is a common reason for intensive care unit (ICU) admission and is associated with prolonged hospital stays and high morbidity and mortality rates. The Atlanta classification differentiates mild, moderate, and severe acute pancreatitis, and each of these categories correlates with morbidity and mortality. Mortality remains high, between 10% and 39%, in severe and moderately severe acute pancreatitis. After the first week, about 30% of patients with necrotizing pancreatitis develop infected pancreatic necrosis (IPN). IPN is a risk factor for mortality.The treatment of IPN combines antibiotics with interventions to remove the infected intra-abdominal material, preferably using minimally invasive techniques such as percutaneous and endoscopic drainage, which have been proven beneficial. In several studies biological markers such as procalcitonin and interleukin 8 were effective in predicting IPN. However, few clinical risk factors for IPN have been reported. Identifying risk factors may help to improve standardized strategies for early diagnosis and treatment, and then patients outcome. Our primary objective was to identify risk factors for IPN in patients admitted to the ICU for acute pancreatitis. Our secondary objective was to describe the management and outcomes of IPN

DETAILED DESCRIPTION:
Using electronic patient data monitoring systems, the investigators reviewed all patients with a diagnosis of acute necrotizing pancreatitis admitted to digestive liver disease unity or ICUs at the Nantes University Hospital, from January 1, 2012, to december 31, 2015. For enrolled patients, general clinical characteristics were collected. Patients were categorized into two groups according to the development of an infected pancreatic necrosis (highly suspected or proven), and the differences of these characteristics between two groups were evaluated. Potential risk factors were collected and studied by using multiple logistic regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age >18 years) with acute necrotizing pancreatitis admitted in an ICU between January 2012 and December 2015 for moderately severe or severe acute pancreatitis were included.
* Organ failure that resolves within 48 h (transient organ failure) and/or local or systemic complications without persistent organ failure or persistent organ failure (>48 h)

Exclusion Criteria:

* mild acute pancreatitis, defined as no organ failure or local complication (No necrosis or peri-pancreatic collection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with acute necrotizing pancreatitis admitted in an ICU between January 2012 and December 2015 for moderately severe or severe acute pancreatitis
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Risk factors of infected pancreatic necrosis | 4 months
  Potential risk factors included patient demographics, disease severity, complications, morphology on CT, and details of the drainage procedure. Univariate analyses examined potential risk factors on outcome (catheter drainage failure). Then, using multiple logistic regression analysis, factors achieving P≤0.1 in univariate analyses were entered into the model predicting the risk of catheter drainage failure

SECONDARY OUTCOMES:
Risk factors of mortality | 4 months
  Potential risk factors included patient demographics, disease severity, complications, morphology on CT, and details of the drainage procedure. Univariate analyses examined potential risk factors on outcome (mortality). Then, using multiple logistic regression analysis, factors achieving P≤0.1 in univariate analyses were entered into the model predicting the risk of non-survival

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Garret, MD, Principal Investigator — Nantes CHU

REFERENCES:
- [Derived] Garret C, Canet E, Corvec S, Boutoille D, Peron M, Archambeaud I, Le Thuaut A, Lascarrou JB, Douane F, Lerhun M, Regenet N, Coron E, Reignier J. Impact of prior antibiotics on infected pancreatic necrosis microbiology in ICU patients: a retrospective cohort study. Ann Intensive Care. 2020 Jun 15;10(1):82. doi: 10.1186/s13613-020-00698-0. PMID 32542577